CLINICAL TRIAL: NCT06094465
Title: Learning Curve of Robotic Pancreatoduodenectomy for Surgeons With Extensive Laparoscopic Pancreatoduodenectomy Experience
Brief Title: Learning Curve of Robotic Pancreatoduodenectomy
Status: Completed | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RPD
Record Dates: First submitted 2023-10-16; First posted 2023-10-23 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Pancreaticoduodenectomy
Keywords: robotic pancreaticoduodenctomy; learning curve

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- learning phase: According to the CUSUM curve, the phase before the peak of the curve is defined as the learning phase.
  Interventions: Other: Different phase of the learning curve of RPD
- proficiency phase: According to the CUSUM curve, the phase after the peak of the curve is defined as the learning phase.
  Interventions: Other: Different phase of the learning curve of RPD

INTERVENTIONS:
Other: Different phase of the learning curve of RPD — Different phases of the learning curve of RPD (learning phase or proficiency phase)

SUMMARY:
A few reports were focused on the RPD learning curve for surgeons with extensive experience in LPD. Therefore, this study aimed to investigate the number of cases required for such surgeons to overcome the learning curve for RPD and to analyze the impact of different phases of the learning curve on perioperative outcomes.

DETAILED DESCRIPTION:
With the development of robotic surgery systems, their unique advantages over traditional laparoscopic surgery systems, such as a three-dimensional 10-fold magnified view, seven degrees of freedom for flexible wrist movements, tremor filtering, and good ergonomic design, have significantly improved the precision and quality of surgery. The literature has reported that, compared with the laparoscopic surgery system, the robotic surgery system can reduce intraoperative blood loss and the conversion rate to laparotomy, in addition to the dissection of more lymph nodes. Therefore, robotic surgery has become increasingly popular. As the economy develops and surgeons gain more experience in LPD, many are shifting their focus to robotic pancreatoduodenectomy after mastering laparoscopic techniques. There are a few reports on the RPD learning curve for surgeons with extensive experience in LPD. Therefore, this study aimed to investigate the number of cases required for such surgeons to overcome the learning curve for RPD and to analyze the impact of different phases of the learning curve on perioperative outcomes.

ELIGIBILITY:
Inclusion Criteria:

patients who received robotic pancreaticoduodenectomy

Exclusion Criteria:

patients who did not receive robotic pancreaticoduodenectomy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: From April 2020 to October 2022, consecutive patients with RPD performed for benign or malignant lesions at Peking Union Medical College Hospital
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
Intraoperative operation time | the data was recorded and collected at the end of the surgery
  Intraoperative operation time, defined as the duration from the skin incision to abdominal closure
Intraoperative blood loss | the data was recorded and collected at the end of the surgery
  Intraoperative blood loss
Conversion to laparotomy | The data was recorded and collected at the end of the surgery
  Conversion to laparotomy
Postoperative complications | up to 3 months after surgery
  Postoperative pancreatic fistula; hemorrhage, abdominal infection, reoperation

CONTACTS AND LOCATIONS:
Overall Officials: Menghua Dai, MD, Study Chair — Peking Union Medical College Hospital
Locations (1):
- Department of General Surgery, Peking Union Medical College Hospital (PUMCH), Peking Union Medical College and Chinese Academy of Medical Sciences, Beijing, China, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Strobel O, Neoptolemos J, Jager D, Buchler MW. Optimizing the outcomes of pancreatic cancer surgery. Nat Rev Clin Oncol. 2019 Jan;16(1):11-26. doi: 10.1038/s41571-018-0112-1. PMID 30341417
- [Result] Gagner M, Pomp A. Laparoscopic pylorus-preserving pancreatoduodenectomy. Surg Endosc. 1994 May;8(5):408-10. doi: 10.1007/BF00642443. PMID 7915434
- [Result] Zhang H, Wu X, Zhu F, Shen M, Tian R, Shi C, Wang X, Xiao G, Guo X, Wang M, Qin R. Systematic review and meta-analysis of minimally invasive versus open approach for pancreaticoduodenectomy. Surg Endosc. 2016 Dec;30(12):5173-5184. doi: 10.1007/s00464-016-4864-3. Epub 2016 Mar 22. PMID 27005287
- [Result] Nickel F, Haney CM, Kowalewski KF, Probst P, Limen EF, Kalkum E, Diener MK, Strobel O, Muller-Stich BP, Hackert T. Laparoscopic Versus Open Pancreaticoduodenectomy: A Systematic Review and Meta-analysis of Randomized Controlled Trials. Ann Surg. 2020 Jan;271(1):54-66. doi: 10.1097/SLA.0000000000003309. PMID 30973388
- [Result] Wang M, Li D, Chen R, Huang X, Li J, Liu Y, Liu J, Cheng W, Chen X, Zhao W, Li J, Tan Z, Huang H, Li D, Zhu F, Qin T, Ma J, Yu G, Zhou B, Zheng S, Tang Y, Han W, Meng L, Ke J, Feng F, Chen B, Yin X, Chen W, Ma H, Xu J, Liu Y, Lin R, Dong Y, Yu Y, Liu J, Zhang H, Qin R; Minimally Invasive Treatment Group in the Pancreatic Disease Branch of China's International Exchange and Promotion Association for Medicine and Healthcare (MITG-P-CPAM). Laparoscopic versus open pancreatoduodenectomy for pancreatic or periampullary tumours: a multicentre, open-label, randomised controlled trial. Lancet Gastroenterol Hepatol. 2021 Jun;6(6):438-447. doi: 10.1016/S2468-1253(21)00054-6. Epub 2021 Apr 27. PMID 33915091
- [Result] Poves I, Burdio F, Morato O, Iglesias M, Radosevic A, Ilzarbe L, Visa L, Grande L. Comparison of Perioperative Outcomes Between Laparoscopic and Open Approach for Pancreatoduodenectomy: The PADULAP Randomized Controlled Trial. Ann Surg. 2018 Nov;268(5):731-739. doi: 10.1097/SLA.0000000000002893. PMID 30138162
- [Result] Zhang H, Lan X, Peng B, Li B. Is total laparoscopic pancreaticoduodenectomy superior to open procedure? A meta-analysis. World J Gastroenterol. 2019 Oct 7;25(37):5711-5731. doi: 10.3748/wjg.v25.i37.5711. PMID 31602170
- [Result] Kamarajah SK, Gujjuri R, Bundred JR, Hilal MA, White SA. Long-term survival after minimally invasive resection versus open pancreaticoduodenectomy for periampullary cancers: a systematic review, meta-analysis and meta-regression. HPB (Oxford). 2021 Feb;23(2):197-205. doi: 10.1016/j.hpb.2020.09.023. Epub 2020 Oct 16. PMID 33077373
- [Result] Kawka M, Gall TMH, Hand F, Nazarian S, Cunningham D, Nicol D, Jiao LR. The influence of procedural volume on short-term outcomes for robotic pancreatoduodenectomy-a cohort study and a learning curve analysis. Surg Endosc. 2023 Jun;37(6):4719-4727. doi: 10.1007/s00464-023-09941-8. Epub 2023 Mar 8. PMID 36890417
- [Result] Boone BA, Zenati M, Hogg ME, Steve J, Moser AJ, Bartlett DL, Zeh HJ, Zureikat AH. Assessment of quality outcomes for robotic pancreaticoduodenectomy: identification of the learning curve. JAMA Surg. 2015 May;150(5):416-22. doi: 10.1001/jamasurg.2015.17. PMID 25761143